CLINICAL TRIAL: NCT03684512
Title: Individual and Family-based Approaches to Increase Physical Activity in Adolescents With IDD
Brief Title: Promotion of Physical Activity in Adolescents With Intellectual and Developmental Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00140784; R01HD094704 (NIH)
Record Dates: First submitted 2018-09-24; First posted 2018-09-25 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Adolescent Behavior; Intellectual Disability; Down Syndrome; Physical Activity
MeSH Terms: conditions — Adolescent Behavior; Intellectual Disability; Down Syndrome; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adolescent Only (Experimental): Remote based physical activity intervention delivered to adolescents only. Adolescents will be asked to attend weekly group exercise sessions, individual support sessions, and monitor their daily physical activity.
  Interventions: Behavioral: Group Exercise Sessions; Behavioral: Individual Support Sessions
- Adolescent and Parent (Active Comparator): Remote based physical activity intervention delivered to adolescents and their parent. Adolescents and a parent will be asked to attend weekly group exercise sessions, individual support sessions, and monitor their daily physical activity. Parents will have access to a Parent Facebook group.
  Interventions: Behavioral: Group Exercise Sessions; Behavioral: Individual Support Sessions; Behavioral: Facebook Group

INTERVENTIONS:
Behavioral: Group Exercise Sessions — Remote exercise sessions delivered over group video conference
Behavioral: Individual Support Sessions — Individual education/support/feedback sessions delivered over video chat
Behavioral: Facebook Group — Facebook group for parents to provide additional support and education
  Arms: Adolescent and Parent

SUMMARY:
The objective of this study is to compare the effect of two strategies to increase MVPA in adolescents with intellectual and developmental disabilities (IDD): a single level intervention delivered to the adolescent only, and a multi-level intervention delivered to both the adolescent and a parent .

DETAILED DESCRIPTION:
We will study adolescents with mild to moderate IDD. Each participant will have 1 designated parent who supports the participant during the physical activity (PA) intervention and in the adolescent and parent arm does the physical activity with the participant. Approximately 29 participants/yr. over 4 yrs. will be randomized in a 1:1 allocation to a remote group-based program of MVPA delivered to the adolescent (AO) or a multi-level intervention delivered to both the adolescent and a parent (A+P). Both interventions will be 12 mos. (6 mos. active intervention, 6 mos. maintenance intervention) with a 6 mos. no-contact follow-up targeted to increase MVPA to the recommended 60 min/d. Both intervention will include real-time MVPA sessions delivered to groups of 5-7 adolescents in their homes using video conferencing software (ZoomTM) with homework assignments designed to increase MVPA on the non-group session days. Parents of adolescents in the A+P group will be asked to participate in the group video MVPA sessions and homework activity, and to attend sessions (0-6 mos. 2 session/mo.; 7-12 mos. 1 session/mo.) with their adolescent and the health coach designed to educate/support parents regarding the role of MVPA in health and function and strategies for increasing MVPA and decreasing sedentary time in both their adolescent and themselves. All participants will monitor their daily PA using a Fitbit wireless activity tracker.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate IDD (IQ of 74-40).
* Sufficient functional ability to understand directions, communicate preferences, wants, and needs through spoken language.
* Living at home with a parent or guardian who is willing to participate in the intervention, with no plans to change this living situation and/or to leave the study area in the next 18 mos.
* Wireless internet access in the home.

Exclusion Criteria:

* Unable to participate in moderate to vigorous physical activity (MVPA).
* Pregnancy during the previous 6 mos., currently lactating, or planned pregnancy in the following 18 mos.
* Unwilling to be randomized.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren T Ptomey, Principal Investigator — University of Kansas; Joseph Donnelly, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas, Lawrence, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ptomey LT, Washburn RA, Lee J, Sherman JR, Rice AM, Danon JC, White DA, Szabo-Reed AN, Helsel BC, Donnelly JE. An Individual versus Parent Supported Physical Activity Intervention in Adolescents with Intellectual Disabilities. Med Sci Sports Exerc. 2024 Dec 1;56(12):2256-2266. doi: 10.1249/MSS.0000000000003515. Epub 2024 Jul 4. PMID 38967389
- [Derived] Ptomey LT, Washburn RA, Lee J, Greene JL, Szabo-Reed AN, Sherman JR, Danon JC, Osborne LN, Little TD, Donnelly JE. Individual and family-based approaches to increase physical activity in adolescents with intellectual and developmental disabilities: Rationale and design for an 18 month randomized trial. Contemp Clin Trials. 2019 Sep;84:105817. doi: 10.1016/j.cct.2019.105817. Epub 2019 Jul 22. PMID 31344519

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Dyads of adolescents with intellectual disabilities and a parent.
Groups:
- Adolescent and Parent (A+P): Remote based physical activity intervention delivered to adolescents and their parent. Adolescents and a parent will be asked to attend weekly group exercise sessions, individual support sessions, and monitor their daily physical activity. Parents will have access to a Parent Facebook group.
  Group Exercise Sessions: Remote exercise sessions delivered over group video conference
  Individual Support Sessions: Individual education/support/feedback sessions delivered over video chat
  Facebook Group: Facebook group for parents to provide additional support and education
- Adolescent Only (AO): Remote based physical activity intervention delivered to adolescents only. Adolescents will be asked to attend weekly group exercise sessions, individual support sessions, and monitor their daily physical activity.
  Group Exercise Sessions: Remote exercise sessions delivered over group video conference
  Individual Support Sessions: Individual education/support/feedback sessions delivered over video chat
Period: Overall Study
Arm/Group | Adolescent and Parent (A+P) | Adolescent Only (AO)
Started | 57 (57 adolescents with intellectual disabilities and 55 parents of adolescents with intellectual disabilities were enrolled. 2 parents had multiple children who enrolled in the intervention together.) | 59 (59 adolescents with intellectual disabilities and 57 parents of adolescents with intellectual disabilities were enrolled. 2 parents had multiple children who enrolled in the intervention together.)
Completed 6 Months | 47 (47 adolescents with intellectual disabilities and 45 parents of adolescents with intellectual disabilities completed the 6 month intervention. 2 parents had multiple children who enrolled in the intervention together and remained in the study at 6 months.) | 54 (54 adolescents with intellectual disabilities and 52 parents of adolescents with intellectual disabilities completed the 6 month intervention. 2 parents had multiple children who enrolled in the intervention together and remained in the study at 6 months.)
Completed 12 Month Active Intervention | 40 (40 adolescents with intellectual disabilities and 38 parents of adolescents with intellectual disabilities completed the12 month intervention. 2 parents had multiple children who enrolled in the intervention together and completed the 12 month intervention.) | 48 (48 adolescents with intellectual disabilities and 46 parents of adolescents with intellectual disabilities completed the12 month intervention. 2 parents had multiple children who enrolled in the intervention together and completed the 12 month intervention.)
Completed | 37 (37 adolescents with intellectual disabilities and 35 parents of adolescents with intellectual disabilities completed the 18 month intervention. 2 parents had multiple children who enrolled in the intervention together and remained in the study until completion.) | 45 (45 adolescents with intellectual disabilities and 43 parents of adolescents with intellectual disabilities completed the 18 month intervention. 2 parents had multiple children who enrolled in the intervention together and remained in the study until completion.)
Not Completed | 20 | 14

BASELINE CHARACTERISTICS:
Population: Participants were adolescents with an intellectual disability and a parent. Note 4 parents (AO: 2, A+P: 2) had 2 children who enrolled in the study together.
Groups:
- Adolescent Only (AO): Adolescents: Remote based physical activity intervention delivered to adolescents only. Adolescents will be asked to attend weekly group exercise sessions and monitor their daily physical activity.
  Group Exercise Sessions: Remote exercise sessions delivered over group video conference
- Adolescent Only (AO): Parents: Parents had adolescents who were randomized to the AO intervention. Parents were not asked to do anything in the intervention.
- Adolescent and Parent (A+P): Adolescents: Remote based physical activity intervention delivered to adolescents and their parent. Adolescents and a parent will be asked to attend weekly group exercise sessions, individual support sessions, and monitor their daily physical activity. Parents will have access to a Parent Facebook group.
  Group Exercise Sessions: Remote exercise sessions delivered over group video conference
  Individual Support Sessions: Individual education/support/feedback sessions delivered over video chat
  Facebook Group: Facebook group for parents to provide additional support and education
- Adolescent and Parent (A+P): Parents: Parents had adolescents who were randomized to the A+P intervention. Parents were asked to attend weekly group exercise session, individual support sessions and had access to a parent facebook group.
  Group Exercise Sessions: Remote exercise sessions delivered over group video conference
  Individual Support Sessions: Individual education/support/feedback sessions delivered over video chat
  Facebook Group: Facebook group for parents to provide additional support and education
- Total: Total of all reporting groups
Arm/Group | Adolescent Only (AO): Adolescents | Adolescent Only (AO): Parents | Adolescent and Parent (A+P): Adolescents | Adolescent and Parent (A+P): Parents | Total
Number analyzed (Participants) | 59 | 57 | 57 | 55 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (3.1) | 47.7 (7.45) | 15.6 (2.9) | 48.6 (7.05) | 31.8 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 52 | 29 | 51 | 163
  Male | 28 | 5 | 28 | 4 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 5 | 3 | 15
  Not Hispanic or Latino | 55 | 54 | 52 | 52 | 213
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 6 | 7 | 4 | 4 | 21
  White | 43 | 46 | 45 | 48 | 182
  More than one race | 7 | 1 | 8 | 3 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Moderate To Vigorous Physical Activity [Mean (Standard Deviation); unit: minutes per day] — Population: For participants in which valid accelerometer data was obtained.
  minutes per day
    number analyzed (Participants) | 52 | 51 | 44 | 47 | 194
    (all) | 22.15 (29.17) | 17.67 (18.02) | 17.01 (15.61) | 16.96 (18.30) | 19.83 (20.95)

OUTCOME MEASURES:

1. Primary Outcome: Change in Adolescent Physical Activity From Baseline to 6 Months
Description: Moderate to vigorous physical activity was assessed using an ActiGraph accelerometer worn during waking hours for 7 consecutive days, with the exception of bathing, and swimming. Data were considered valid if they wore the accelerometer for at least 8 hours on 3 days, including 1 weekend day.
Time Frame: Change from baseline to 6 months
Population: Adolescents who had valid accelerometer data at both baseline and 6 months
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Adolescent Only (AO) | Adolescent and Parent (A+P)
Number analyzed (Participants) | 42 | 31
minutes per day | -3.2 (14.8) | -0.6 (12.5)

2. Secondary Outcome: Change in Adolescent Moderate to Vigorous Physical Activity From Baseline to 18 Months
Description: as for outcome 1
Time Frame: Change from baseline to 18 months
Population: Adolescents who had valid accelerometer data at both baseline and 18 months
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Adolescent Only (AO) | Adolescent and Parent (A+P)
Number analyzed (Participants) | 32 | 23
minutes per day | -1.5 (28.5) | 7.6 (21.8)

3. Secondary Outcome: Change in Parent Physical Activity
Description: Moderate to Vigorous Physical Activity in parents of participants will be assessed at baseline, 3, 6, 12, and 18 months using an ActiGraph accelerometer over 7 days
Time Frame: Change from baseline to 18 months
Reporting Status: Not Posted

4. Secondary Outcome: Change in Sedentary Time
Description: Sedentary Time in adolescents with IDD will be assessed at baseline, 3, 6, 12, and 18 months, using an ActiGraph accelerometer over 7 days.
Time Frame: Change from baseline to 18 months
Reporting Status: Not Posted

5. Secondary Outcome: Change in Parent Sedentary Time
Description: Sedentary Time in parents of participants will be assessed at baseline, 3, 6, 12, and 18 months, using an ActiGraph accelerometer over 7 days.
Time Frame: Change from baseline to 18 months
Reporting Status: Not Posted

6. Secondary Outcome: Change in Cardiovascular Fitness
Description: Cardiovascular fitness will be assessed by treadmill at baseline, 3, 6, 12, and 18 months
Time Frame: Change from baseline to 18 months
Reporting Status: Not Posted

7. Secondary Outcome: Change in Muscular Strength
Description: Assessed at baseline, 6, 12, and 18 months by chest press and leg press
Time Frame: Change from baseline to 18 months
Reporting Status: Not Posted

8. Secondary Outcome: Change in Motor Ability
Description: Assessed by the Gross Motor Quotient and Percentile obtained from Test of Gross Motor Development-second edition
Time Frame: Change from baseline to 18 months
Reporting Status: Not Posted

9. Secondary Outcome: Change in Quality of Life
Description: Assessed a using the PedsQL 4.0 Generic Core Scale designed to measure health-related quality of life in healthy children and adolescents and in those with chronic health conditions
Time Frame: Change from baseline to 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 18 months
Description: Adverse events were only collected from the adolescent.
Arm/Group | Adolescent Only | Adolescent and Parent
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/57
Serious Adverse Events (participants affected / at risk) | 2/59 | 1/57
Other Adverse Events (participants affected / at risk) | 1/59 | 2/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adolescent Only (N=59) | Adolescent and Parent (N=57)
COVID 19 Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Pancreatitis (Endocrine disorders) | 1 (1) | 0
Tubulointerstitial Nephritis (Renal and urinary disorders) | 1 (2) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adolescent Only (N=59) | Adolescent and Parent (N=57)
Rash from Fitbit Watch (Product Issues) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT03684512/Prot_SAP_000.pdf